CLINICAL TRIAL: NCT04523467
Title: A Multicentre Randomized Controlled Study of Anti-angiogenic Targeted Drugs Combined With Ginsenoside Rg3 to Improve the Efficacy of Transcatheter Arterial Chemoembolization (TACE) in the Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Anti-angiogenic Targeted Drugs Plus Rg3 to Improve the Efficacy of TACE for Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, MD, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2020-K-009
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — ginsenoside Rg3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined group (Experimental): Anti-angiogenic targeted drug + Rg3 + TACE
  Interventions: Drug: Anti-angiogenic Targeted Drugs; Drug: Ginsenoside Rg3; Procedure: TACE
- Single group (Active Comparator): TACE alone
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: Anti-angiogenic Targeted Drugs — A tyrosine kinase inhibitor inhibits vascular endothelial growth factor (VEGF) receptors 1-3, showed efficacy in hepatocellular carcinoma
  Other Names: TKI Drugs
  Arms: Combined group
Drug: Ginsenoside Rg3 — An active ingredient extracted from ginseng leachate, which can restrain angiogenesis and reduce the expression of programmed cell death ligand 1 (PD-L1) on the tumor cell surface and block the binding of programmed cell death 1 (PD-1) and PD-L1
  Other Names: Rg3
  Arms: Combined group
Procedure: TACE — A specific type of chemoembolization that blocks the hepatic artery to treat liver cancer

SUMMARY:
The aim of this study is to compare the efficacy and safety of transcatheter arterial chemoembolization (TACE) combined with the anti-angiogenic targeted drugs and ginsenoside Rg3 versus TACE alone in patients with unresectable Barcelona Clinic Liver Cancer (BCLC) stage B/C hepatocellular carcinoma (HCC), who has normal liver function and no extrahepatic metastasis.

DETAILED DESCRIPTION:
TACE is widely used in patients with unresectable HCC, which has been proved to significantly improve the survival time by the results from some randomized controlled studies and meta-analyses. However, due to the different blood supply characteristics and biological heterogeneity in HCC nodules, the therapeutic effect of TACE is limited, and which is still considered as a non-radical treatment. Furthermore, vascular embolization by TACE may result in hypoxia in tumor tissue, which will induce increased secretion of angiogenic factors such as vascular endothelial growth factor (VEGF) and tumor angiogenesis, promote proliferation of residual tumor cells, and enhance tumor invasive and metastasis. Accordingly, the effectiveness of TACE is still unsatisfying as a single treatment for HCC.

Both anti-angiogenic targeted drugs and ginsenoside Rg3 have showed synergistic effect with TACE in patients with unresectable HCC. The purpose of this trial is to evaluate the efficacy and safety of the combination of anti-angiogenic targeted drugs and ginsenoside Rg3 plus TACE comparing to TACE alone in patients with unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75
2. Unresectable HCC patients clinically diagnosed or confirmed by histopathology and/or cytology according to Guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2019 edition);
3. At least one measurable lesion (according to mRECIST);
4. BCLC stage B or C (China Liver Cancer Staging [CNLC] IIa, IIb and IIIa);
5. The maximum diameter of a single lesion ≤10cm; No more than 10 lesions; or combined with portal vein thrombus (PVTT) type I and II (Cheng's classification);
6. Child-pugh score <7;
7. Eastern Cooperative Oncology Group (ECOG) PS 0-1;

Exclusion Criteria:

1. Mixed hepatocellular carcinoma and intrahepatic cholangiocarcinoma (HCC-ICC) confirmed by pathology;
2. Extrahepatic metastasis;
3. Previously received hepatectomy, liver transplantation, interventional therapy, ablative therapy and other local therapies for HCC;
4. PVTT type III/IV (Cheng's classification), major hepatic vein invasion or primary to secondary bile duct invasion;
5. A history of gastrointestinal bleeding or a definite tendency of gastrointestinal bleeding in the past 4 weeks;
6. Cardiovascular diseases with significant clinical significance;
7. Active infection;
8. Other significant clinical and laboratory abnormalities that investigators believe affect safety evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  the time from randomization to documented progression

SECONDARY OUTCOMES:
Time to TACE untreated progression | Up to 2 years
  the time from randomization to TACE untreatable progression
Objective response rate | Up to 2 years
  The proportion of patients whose tumor volume has decreased to a predetermined value
Overall survival | Up to 2 years
  The time period from the randomization of the patient to the death event due to any reason
Adverse events | Up to 2 years
  The severity of adverse events will be evaluated according to the NCI CTCAE 5.0 standard the severity of adverse events will be evaluated according to the NCI CTCAE 5.0 standard the severity of adverse events will be evaluated according to the NCI CTCAE 5.0 standard

OTHER OUTCOMES:
Conversion rate | Up to 2 years
  The proportion of patients whose tumor has changed from unresectable to resectable after Intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China